CLINICAL TRIAL: NCT05338281
Title: Negative Pressure Wound Therapy for Abdominal Incisions in DIEP Reconstructions: A RCT
Brief Title: NPWT for Abdominal Incisions in DIEP Reconstructions: A RCT
Acronym: NPWTinDIEP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study details changed, new Trial Registration process begun for modified protocol
Sponsor: Western University, Canada (Other)
Collaborators: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Tanya DeLyzer, Principal Investigator, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 120134
Record Dates: First submitted 2022-04-13; First posted 2022-04-21 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Surgical Site Infection; Wound Dehiscence
Keywords: DIEP; Negative Pressure Wound Therapy; Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms; Surgical Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Negative Pressure Wound Therapy (Experimental): This group will receive the usual care of the abdominal donor wound following DIEP flap-based breast reconstruction surgery, AND the negative pressure wound therapy. The Prevena™ Incision Management System will be placed at the abdominal flap donor site after incision is closed. The Prevena™ will remain for up to 5 days, or until patient is discharged from the hospital.
  Interventions: Device: Negative Pressure Wound Therapy
- Standard Dressing (Active Comparator): This group will receive the usual care of the abdominal donor wound following DIEP flap-based breast reconstruction surgery, and standard dressing which will be composed of gauze, secured with paper tape.
  Interventions: Device: Negative Pressure Wound Therapy

INTERVENTIONS:
Device: Negative Pressure Wound Therapy — The negative pressure wound therapy will be placed in addition to usual care of the abdominal donor site, such as closure with resorbable sutures, drain placements.
  Other Names: Prevena™ Incision Management System

SUMMARY:
The current study is a single center randomized control trial that will examine the effect of closed incision negative pressure wound therapy (ciNPT) versus conventional dressing on abdominal incision in a deep inferior epigastric perforator (DIEP) flap based reconstruction. Patients will be followed by 30 days post-operatively to compare outcomes including the rate of surgical site infection, seroma, and the scar quality.

DETAILED DESCRIPTION:
The current study will examine the effect of closed incision negative pressure wound therapy on DIEP flap donor site. A total of 520 patients who are candidates for DIEP flap-based breast reconstruction will be included in this study, and randomly divided into the two groups. Those with contraindications to ciNPT will be excluded. The surgical consultation and procedure will be conducted same for both groups. Patients will be followed by 30 days post-operatively. Outcome measures will include incidence of surgical site infection, wound dehiscence, seroma, hematoma, delayed wound healing, and surgical scar quality.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing either immediate, or delayed reconstruction of the breast following mastectomy
* Patients going either unilateral or bilateral reconstruction

Exclusion Criteria:

* Patients who are not candidates for DIEP flap based breast reconstruction, such as those with insufficient abdominal tissue, or unfit for the surgery will be excluded from this study. -
* Patients who have contraindications to the ciNPT
* Patients who have pre-existing conditions that may confound results such as bleeding disorder or therapeutic anticoagulation will be excluded from the study.
* Patients who do not want to carry an additional canister from the ciNPT during the initial recovery phase will be excluded from the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative Surgical Site Infection (SSI) | 30 days after operation
  The post-operative SSI at the abdomen will be determined following the Center for Disease Control (CDC) criteria. This includes one or more of the following:
  1. Purulent drainage from the incision, 2. Organisms identified from an aseptically-obtained specimen 3. Superficial incision with one of the following signs or symptoms localized pain or tenderness; localized swelling; erythema; or heat.
  d. Diagnosis of a superficial incisional SSI by a physician or designee

SECONDARY OUTCOMES:
The rate of seroma diagnosis | 30 days after operation
  The diagnosis of seroma will be completed by clinical exam and/or diagnostic imaging such as ultrasound or computed tomography.
The rate of hematoma diagnosis | 30 days after operation
  The diagnosis of hematoma will be completed by clinical exam and/or diagnostic imaging such as ultrasound or computed tomography.
The rate of wound dehiscence | 30 days after operation
  The diagnosis of wound dehiscence will be made by clinical exam.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya DeLyzer, MD, FRCSC, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No